CLINICAL TRIAL: NCT06887699
Title: A Randomized Clinical Trial Investigating the Impact of Artificial Intelligence Electrocardiography on Occlusion Myocardial Infarction Management Under the Value-Based Payment System
Brief Title: The Impact of Artificial Intelligence Electrocardiography on Occlusion Myocardial Infarction Management Under the Value-Based Payment System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Chin Lin, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: A202505035
Record Dates: First submitted 2025-03-04; First posted 2025-03-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: OMI - Occlusion Myocardial Infarction; Artificial Intelligence (AI); Electrocardiogram; Cost-effectiveness Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-ECG P4P program (Experimental): AI-ECG-assisted detection of OMI within the P4P program. The AI-ECG system will conduct a real-time analysis of the ECG. When the system identifies potential OMI cases, it will immediately send short message service notifications to the on-duty cardiologists. This will enable the cardiologists to promptly review and confirm the diagnosis.
  Interventions: Other: AI-ECG P4P program
- Standard of care (No Intervention): Potential OMI patients will be initially assessed by frontline physicians. If OMI is suspected, the frontline physicians will promptly notify the on-duty cardiologists, who will then review the case for confirmation.

INTERVENTIONS:
Other: AI-ECG P4P program — The AI-ECG system will conduct a real-time analysis of the ECG. When the system identifies potential OMI cases, it will immediately send short message service notifications to the on-duty cardiologists. This will enable the cardiologists to promptly review and confirm the diagnosis.
  Arms: AI-ECG P4P program

SUMMARY:
This trial will prospectively evaluate the impact of integrating AI-ECG within the pay-for-performance program on improving the diagnosis, treatment, and clinical outcomes of occlusion myocardial infarction patients by promoting accurate and timely diagnoses through financial incentives.

DETAILED DESCRIPTION:
The investigators have developed an AI-ECG system that provides real-time notifications for patients with potential occlusion myocardial infarction. This AI algorithm is seamlessly integrated into the Hospital Information System, allowing for the automatic generation of reports whenever an ECG is performed. The purpose of this study is to evaluate the impact of AI-ECG on the timely diagnosis of STEMI, including patients' outcomes and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the emergency department
* Patients received at least 1 ECG examination.

Exclusion Criteria:

* The patients received ECG at the period of inactive AI-ECG system.
* Patients with a history of coronary angiography within the past 3 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212000 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
D-to-W time (Door to Wire Time) | From the start of the emergency visit to the following 48 hours.
  Door-to-wire time refers to the duration from a patient's arrival at the emergency department (ED) to the successful placement of a wire into the coronary artery during a primary percutaneous coronary intervention (PPCI) procedure.
Cost Outcome Measure | From the start of the emergency visit to 90 days post-discharge.
  Total expenditures, from the start of the emergency visit to 90 days post-discharge (in USD), for comparison between the intervention and control groups, based on records from NHI (National Health Insurance) claims data.

SECONDARY OUTCOMES:
Door-to-Wire time less than 90 minutes | 48 hours
  The proportion of patients achieving a Door-to-Wire time of less than 90 minutes in the intervention group compared to the control group. The intervention and control groups' door-to-wire time will be compared. Door-to-wire time is defined as the duration from the first ECG to the successful placement of the wire during PPCI for OMI patients in the emergent department.
In-hospital all-cause Mortality Rate | 90-day follow
  The proportion of patients who die from any cause, regardless of the underlying condition, during hospitalization.
In-hospital cardiac death | 90-day follow
  The proportion of patients who die from cardiovascular-related causes during hospitalization.
Length of ICU | 90-day follow
  Comparison of length of ICU between the intervention and control groups.
Length of hospitalization | 90-day follow
  Comparison of length of hospitalization between the intervention and control groups.
Cardiovascular events | 90-day follow
  Composite cardiovascular events (Non-fatal MI + Non-fatal stroke + CV Death) The rate of composite cardiovascular events within 90 days.
Non-fatal MI | 90-day follow
  The rate of non-fatal MI within 90-days.
Non-fatal stroke (Ischemic stroke + Hemorrhagic stroke) | 90-day follow
  The rate of non-fatal strokes (both ischemic and hemorrhagic) within 90-days.
Cardiac Death | 90-day follow
  The proportion of patients who die from cardiovascular-related causes within 90-days.
Ischemic stroke | 90-day follow
  The incidence of ischemic stroke.
Hemorrhagic stroke | 90-day follow
  The incidence of hemorrhagic stroke.
All-cause mortality | 90-day follow
  The proportion of patients who die from any cause within 90-days.
Coronary artery bypass grafting (CABG) | 90-day follow
  The rate of patients who undergo coronary artery bypass surgery (CABG) within 90-days following OMI treatment.
Heart failure admission | 90-day follow
  The rate of hospital admissions for heart failure within 90-days following OMI treatment.
Re-hospitalization (from any cause) | 90-day follow
  The rate of readmission to the hospital within 90-days of discharge.

OTHER OUTCOMES:
Emergent CAG without PCI | From the start of the emergency visit to the following 48 hours.
  The number of patients who received emergent coronary angiograms without lesions need intervention.
Procedure related vascular complications | From the start of the emergency visit to the following 48 hours.
  The number of patients who received a procedure with vascular complications.
Contrast-induced acute kidney injury | 90-day follow
  The number of patients who received a procedure with contrast-induced acute kidney injury.
Procedure related mortality | 90-day follow
  The proportion of patients who die due to the procedure within 90 days.
In-hospital major bleeding | 90-day follow
  The incidence of in-hospital major bleeding events occurring within 90-days of treatment.
Major bleeding | 90-day follow
  The incidence of major bleeding events occurring within 90-days of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chin Lin, PhD, Principal Investigator — National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No